CLINICAL TRIAL: NCT00730444
Title: Expanded Access Protocol for [123I]mIBG for Patients With Known or Suspected Neuroblastoma
Status: Approved for marketing | Type: Expanded Access
Sponsor: GE Healthcare (Industry)
Responsible Party: Arnold F. jacobson, M.D., PhD./Clinical Project Leader, GE Healthcare Ltd. and its affiliates
Other Study IDs: GE 122-008
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Nuclear medicine; Diagnostic scintigraphy; Known and suspected neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine

INTERVENTIONS:
Drug: Iobenguane I 123 Injection — 1-10 mCi administered intravenously
  Other Names: AdreView

SUMMARY:
GE Healthcare has recently submitted a New Drug Application (NDA) for Iobenguane I 123 Injection ([123I]mIBG (AdreView)) as a diagnostic nuclear imaging agent for the detection of primary or metastatic neuroblastoma and pheochromocytoma. The present protocol establishes an Expanded Access program to provide AdreView to pediatric medical centers and hospitals that treat neuroblastoma patients. AdreView will be provided for use in diagnostic assessment of patients with known or suspected neuroblastoma for whom there is an appropriate clinical indication for [123I]mIBG imaging.

DETAILED DESCRIPTION:
The sponsor will provide [123I]mIBG as a single dose in a ready-to-use vial. All patients greater than or equal to 18 years of age and children with a weight of greater than or equal to 70 kg will receive an intravenous injection of 370 ±10% MBq (333 to 407 MBq [9.0 to 11 mCi]) of [123I]mIBG. Children <16 years of age (with a weight of 8-70 kg) will receive an activity of [123I]mIBG calculated on the basis of a reference activity for an adult scaled to body weight. Each investigator is responsible for obtaining the appropriate thyroid blockade agent and for its administration in accordance with national and local regulations and guidelines. Approximately 24 (± 6) hours following administration of [123I]mIBG all patients will return to the clinic for scintigraphic imaging. Imaging will be performed as per the standard procedures of the investigational site. This should include at a minimum total body planar scintigraphy. Single photon emission computed tomography (SPECT) may be performed following planar scintigraphy, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* The patient has known or suspected neuroblastoma and is undergoing evaluation of disease status (for which a mIBG scintigraphic examination is clinically appropriate).
* The patient is able and willing to comply with study procedures and a signed and dated informed consent is obtained from the patient (or their legal guardian.

Exclusion Criteria:

* The patient uses medications that are known to interfere with [123I]mIBG uptake and these medications cannot be safely withheld for a least 24 hours before study procedures.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Jacobson, MD, Principal Investigator — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States